CLINICAL TRIAL: NCT04708067
Title: "Window of Opportunity" Phase I Trial of Focal Radiotherapy and Bintrafusp Alfa In Patients With Advanced Intrahepatic Cholangiocarcinoma
Brief Title: Hypofractionated Radiation Therapy and Bintrafusp Alfa for the Treatment of Advanced Intrahepatic Cholangiocarcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0899; NCI-2020-13928 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0899 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Intrahepatic Cholangiocarcinoma; Metastatic Intrahepatic Cholangiocarcinoma; Stage III Intrahepatic Cholangiocarcinoma AJCC v8; Stage IIIA Intrahepatic Cholangiocarcinoma AJCC v8; Stage IIIB Intrahepatic Cholangiocarcinoma AJCC v8; Stage IV Intrahepatic Cholangiocarcinoma AJCC v8
MeSH Terms: conditions — Cholangiocarcinoma | interventions — bintrafusp alfa protein, human; Biopsy; Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (hypofractionated radiation, bintrafusp alfa) (Experimental): Patients undergo hypofractionated radiation therapy QD on weekdays (Monday-Friday) for 15 fractions in the absence of disease progression or unacceptable toxicity. Beginning 1 week after completion of radiation therapy, patients receive bintrafusp alfa IV over 1 hour on day 1. Cycles repeat every 14 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bintrafusp Alfa; Procedure: Biopsy; Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Drug: Bintrafusp Alfa — Given IV
  Other Names: Anti-PDL1/TGFb Trap MSB0011359C; M7824; MSB0011359C
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation

SUMMARY:
This phase I trial is to find out the best dose, possible benefits, and/or side effects of hypofractionated radiation therapy and bintrafusp alfa in treating patients with bile duct cancer that has spread to other places in the body (advanced intrahepatic cholangiocarcinoma). Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Immunotherapy with bintrafusp alfa, a bifunctional fusion protein composed of the monoclonal antibody avelumab and TGF-beta, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. The combination of hypofractionated radiation therapy and bintrafusp alfa may help to control intrahepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the safety of bintrafusp alfa in combination with hypofractionated radiation therapy for patients with advanced intrahepatic cholangiocarcinoma and recommend a phase II radiation dose.

SECONDARY OBJECTIVES:

I. To estimate objective response rate, local progression free survival, progression free survival, overall survival with the study regimen.

II. To correlate expression of TGF-beta related pathways with clinical outcomes.

III. To examine intratumoral pharmacodynamic changes in the immune microenvironment using paired biopsies before and after therapy with the study agents.

EXPLORATORY OBJECTIVE:

I. To correlate immune biomarkers from pre- and post-treatment tissue, blood, and stool with clinical study endpoints.

OUTLINE: This is a dose de-escalation study of radiation therapy followed by a dose-expansion study.

Patients undergo hypofractionated radiation therapy once daily (QD) on weekdays (Monday-Friday) for 15 fractions in the absence of disease progression or unacceptable toxicity. Beginning 1 week after completion of radiation therapy, patients receive bintrafusp alfa intravenously (IV) over 1 hour on day 1. Cycles repeat every 14 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be male or female >= 18 years of age
* Patients with histologically or cytologically confirmed intrahepatic cholangiocarcinoma. There must be at least two measurable tumors. One larger mass that will be radiated and a secondary metastatic site that is amenable to biopsies
* Patients must have received at least one standard first-line chemotherapy regimen or have refused chemotherapy
* Patients with measurable disease assessed at baseline by computed tomography (CT) (or magnetic resonance imaging [MRI] where CT is contraindicated) will be entered in this study
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky > 70)
* Leukocytes >= 3,000 cells/mm^3
* Absolute neutrophil count >= 1,500 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin >= 9 g/dl (no blood transfusions within 4 weeks prior to enrollment)
* Total bilirubin < 1.5 x institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x IULN without liver metastasis, =< 5 x IULN for patients with liver metastasis
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of childbearing potential (defined as not post-menopausal for 65 days or no previous surgical sterilization) and fertile men must agree to use adequate contraception for the duration of study participation
* All female patients of childbearing potential (defined as not post-menopausal for 65 days or no previous surgical sterilization) must agree to use adequate birth control during study treatment and for 90 days after the last dose of study drug and have a negative serum pregnancy test at screening
* Fertile males must be willing to employ adequate means of contraception during study treatment and for 3 months after the last dose of study drug
* Male subjects must agree to refrain from sperm donation during the study and for 125 days after the last dose of study drugs
* Ability to read and/or understand the details of the study and provide written evidence of informed consent as approved by Institutional Review Board (IRB)/ Scientific Review Committee (SRC)

Exclusion Criteria:

* Patients who are pregnant or lactating
* Patients with uncontrolled intercurrent illness including symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia and myocardial infarction (MI) within 3 months of initiation of therapy
* Patients with recent bacterial, viral, or fungal infection(s) requiring systemic antibiotic therapy within one month of enrolling
* Patient has undergone major surgery within 4 weeks prior to day 1 of treatment in this study. Diagnostic or minimally invasive surgery (i.e., done to obtain a biopsy for diagnosis without removal of an organ or to place an abdominal spacer) are acceptable at physician discretion
* Patient received radiotherapy, surgery, chemotherapy, or an investigational therapy within 2 weeks prior to study entry weeks
* Patient has serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive an experimental research drug
* Serious psychiatric or medical conditions that could interfere with treatment
* Major bleeding in the last 4 weeks
* Receipt of prior immune checkpoint inhibitors (e.g., anti-CTLA-4, anti-programmed cell death receptor 1, anti-programmed cell death ligand 1 [anti-PD-L1], and any other antibody or drug specifically targeting T-cell costimulation)
* Receiving an immunologically based treatment for any reason, including chronic use of systemic steroid at doses >= 7.5 mg/day prednisone equivalent within 14 days prior to the first dose of study treatment. Use of inhaled or topical steroids or systemic corticosteroids < 7.5 mg is permitted
* Receipt of any anticancer medication in the 21 days prior to receiving the first dose of study medication or any unresolved toxicity (> grade 1) from previous anticancer therapy, except for stable chronic toxicities not expected to resolve, such as peripheral neurotoxicity. Prior treatment with nitrosoureas (e.g., carmustine or lomustine) require a 6-week washout prior to the first dose of study treatment
* Untreated central nervous system (CNS) metastases, or CNS metastases that have progressed (e.g., evidence of new or enlarging CNS metastasis or new neurological symptoms attributable to CNS metastases). Subjects with treated and clinically stable CNS metastases and off all corticosteroids for at least 2 weeks are eligible
* Any active or inactive autoimmune process (e.g. rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease) or who are receiving systemic therapy for an autoimmune or inflammatory disease

  * Note: Exceptions include subjects with vitiligo, hypothyroidism stable on hormone replacement, controlled asthma, type I diabetes, Graves' disease, or Hashimoto's disease, or with medical monitor approval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 60 days
  AEs will be graded according to Common Terminology Criteria for Adverse Events version 5.0. AEs will be summarized by patient incidence rates, therefore, in any tabulation, a patient contributes only once to the count for a given AE preferred term. The number and percentage of patients with any treatment-emergent AE will be summarized for all study patients combined.

SECONDARY OUTCOMES:
Objective response rate | Up to 2 years post-treatment
  Will estimate the objective response rate by Response Evaluation Criteria in Solid Tumors 1.1 criteria separately with appropriate 95% confidence intervals.
Local progression free survival (LPFS) | Up to 12 months post-treatment
  Will estimate the LPFS distributions using the Kaplan-Meier product limit method and report summary measures such as the median value and probabilities at selected times with appropriate 95% confidence intervals.
Progression free survival (PFS) | Up to 12 months post-treatment
  Will estimate the PFS distributions using the Kaplan-Meier product limit method and report summary measures such as the median value and probabilities at selected times with appropriate 95% confidence intervals.
Overall survival (OS) | Up to 12 months post-treatment
  Will estimate the OS distributions using the Kaplan-Meier product limit method and report summary measures such as the median value and probabilities at selected times with appropriate 95% confidence intervals.

OTHER OUTCOMES:
Biomarker analysis | Up to 2 years post-treatment
  Will analyze changes in biomarker expression before and after treatment using a paired t-test if the data are normally distributed, and a Wilcoxon signed rank test if not. Will correlate biomarker expression with clinical benefit using receiver operator characteristics curve analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene J Koay, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MDAndersonCancerCenterWebsite — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT04708067/ICF_000.pdf